CLINICAL TRIAL: NCT05105932
Title: The Study of Regional Lung Ventilation-perfusion by EIT
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking Union Medical College Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: PUMCH-EIT-PE
Record Dates: First submitted 2021-01-28; First posted 2021-11-03 (Actual); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Pulmonary Ventilation; Pulmonary Perfusion
Keywords: EIT; pulmonary perfusion

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- EIT group: patients went through EIT detection
- CTPA group: patients went through CTPA detection

SUMMARY:
This is a prospective observational trial. The purpose of this study is to explore the feasibility of EIT monitoring pulmonary blood flow and the consistency and difference between EIT monitoring pulmonary local ventilation blood flow and SPECT and CTPA monitoring methods

ELIGIBILITY:
Inclusion Criteria:

1. Admission to ICU was less than 72 hours;
2. Age ≥ 18 years old and ≤ 80 years old;
3. Volunteer to participate after communicating with patients' family members;

Exclusion Criteria:

1. The patients with heart implants could not be monitored by EIT;
2. Patients or their families refused to participate in the study;
3. Hypernatremia

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients who need CTPA examination in the Department of nuclear medicine / radiology of Peking Union Medical College Hospital
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-06-01 (Estimated)

PRIMARY OUTCOMES:
Regional pulmonary perfusion by EIT | 1 Day
  Using EIT to measure the regional pulmonary perfusion and calculate ventilation/perfusion ratio
Regional pulmonary perfusion by CTPA | 1 Day
  Using CTPA to measure the regional pulmonary perfusion and calculate ventilation/perfusion ratio

SECONDARY OUTCOMES:
Regional pulmonary ventilation index by EIT | 1 Day
  Regional pulmonary ventilation index by EIT, including GI: global inhomogeneity CoV: center of ventilation, ROI: region of interest

CONTACTS AND LOCATIONS:
Overall Officials: Yun Long, Study Director — Peking Union Medical College Hospital
Locations (1):
- Peking Union Medical College Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided